CLINICAL TRIAL: NCT01536158
Title: Oral Paracetamol Versus Oral Ibuprofen Treatment
Brief Title: Oral Paracetamol Versus Oral Ibuprofen in Management of Patent Ductus Arteriosus in Preterm Infants: A Randomised Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Yekta, Zekai Tahir Burak Maternity and Teaching Hospital, Zekai Tahir Burak Women's Health Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZTB150212
Record Dates: First submitted 2012-02-15; First posted 2012-02-20 (Estimated); Last update posted 2012-12-27 (Estimated); Status verified 2012-12

CONDITIONS: Patent Ductus Arteriosus
Keywords: Patent Ductus Arteriosus; Paracetamol; Ibuprofen; Preterm infant
MeSH Terms: conditions — Ductus Arteriosus, Patent; Premature Birth | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral paracetamol (Active Comparator): Patients will receive oral paracetamol 15 mg/kg per dose every 6 hours.
  Interventions: Drug: Oral paracetamol
- Oral ibuprofen (Active Comparator): Patients will receive oral ibuprofen at an initial dose of 10 mg/kg, followed by 5 mg/kg at 24 and 48 h.
  Interventions: Drug: Oral ibuprofen

INTERVENTIONS:
Drug: Oral paracetamol — Patients will receive oral paracetamol 15 mg/kg per dose every 6 hours for 3 days.
  Other Names: Calpol
  Arms: Oral paracetamol
Drug: Oral ibuprofen — Patients will receive oral ibuprofen at an initial dose of 10 mg/kg, followed by 5 mg/kg at 24 and 48 h.
  Other Names: Pedifen
  Arms: Oral ibuprofen

SUMMARY:
The purpose of this study is to determine whether oral paracetamol or ibuprofen has a better or same efficacy and tolerance in closure of patent ductus arteriosus in preterm infants.

DETAILED DESCRIPTION:
To determine whether oral paracetamol or ibuprofen has a better or same efficacy and tolerance in closure of patent ductus arteriosus in preterm infants.

Eighty preterm infants with patent ductus arteriosus will be enrolled in this prospective-randomized study. Patients will receive oral ibuprofen at an initial dose of 10 mg/kg, followed by 5 mg/kg at 24 and 48 h or oral paracetamol 15 mg/kg per dose every 6 hours.

One of the following echocardiographic criteria of a duct size >1.5 mm, a left atrium-to-aorta ratio >1.5, left-to-right shunting of blood, end diastolic reversal of blood flow in the aorta, or poor cardiac function in addition signs of patent ductus arteriosis determined the need of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight below 1250 gram
* Diagnosed patent ductus arteriosus by Echocardiographic examination

Exclusion Criteria:

* Accompanied other congenital cardiac anomalies
* Urine output of less than 1 ml/kg/h during the preceding 8 h,
* Serum creatinine level >1.6 mg/dl,
* Platelet count <60,000/mm3,
* Liver failure,
* Hyperbilirubinemia requiring exchange transfusion
* Severe intracranial bleeding (Grade III - IV)
* Intestinal abnormality and necrotising enterocolitis

Ages: 2 Days to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2012-02; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Efficacy and Safety of Oral Paracetamol Versus Oral Ibuprofen | Until discharge
  To compare the closure rate of patent ductus arteriosus after oral paracetamol or oral ibuprofen treatment

SECONDARY OUTCOMES:
Long term effects of oral paracetamol versus oral ibuprofen treatment in preterm infants | corrected 36 weeks or until discharge
  Long term effects such as ROP, BPD,IVH, duration of respiratory support and hospitalization are going to be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Yekta Oncel, MD, Principal Investigator — Zekai Tahir Burak Women's Health Research and Education Hospital
Locations (1):
- Zekai Tahir Burak Maternity Teaching Hospital, Division of Neonatology, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Jasani B, Mitra S, Shah PS. Paracetamol (acetaminophen) for patent ductus arteriosus in preterm or low birth weight infants. Cochrane Database Syst Rev. 2022 Dec 15;12(12):CD010061. doi: 10.1002/14651858.CD010061.pub5. PMID 36519620
- [Derived] Oncel MY, Eras Z, Uras N, Canpolat FE, Erdeve O, Oguz SS. Neurodevelopmental Outcomes of Preterm Infants Treated with Oral Paracetamol Versus Ibuprofen for Patent Ductus Arteriosus. Am J Perinatol. 2017 Oct;34(12):1185-1189. doi: 10.1055/s-0037-1601564. Epub 2017 Apr 10. PMID 28395364
- [Derived] Oncel MY, Yurttutan S, Erdeve O, Uras N, Altug N, Oguz SS, Canpolat FE, Dilmen U. Oral paracetamol versus oral ibuprofen in the management of patent ductus arteriosus in preterm infants: a randomized controlled trial. J Pediatr. 2014 Mar;164(3):510-4.e1. doi: 10.1016/j.jpeds.2013.11.008. Epub 2013 Dec 18. PMID 24359938
- See also: Ibuprofen — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0015687271&QV1=IBUPROFEN
- See also: Paracetamol — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0000103902&QV1=PARACETAMOL